CLINICAL TRIAL: NCT04097249
Title: The Contribution and Validity of Infrared Thermography in the Diagnosis of Musculoskeletal Pain
Brief Title: Infrared Thermography for the Diagnosis of Musculoskeletal Pain
Status: Completed | Type: Observational
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Other Study IDs: P15/2015
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Healthy; Pain; Temperature Change, Body
Keywords: Musculoskeletal pain; Delayed Onset Muscle Soreness; Pain sensitivity; Infrared thermography; Referred pain
MeSH Terms: conditions — Pain; Body Temperature Changes; Musculoskeletal Pain; Pain, Referred

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects: Participants free from any pain specific to the upper limb, chronic pain or other disease.

SUMMARY:
This study sought to evaluate the vasomotor response in the pain referral area of healthy individuals, performing the same procedure with and without the experience of delayed onset muscle soreness.

DETAILED DESCRIPTION:
Validity of infrared thermography for properly diagnosing musculoskeletal pain and their clinical applicability is lacking. This study investigates temperature changes on the upper extremity before and after a suprathreshold stimulation (painful stimulus) with a digital algometer over the infraspinatus muscle. The same procedure is performed in two consecutive days, 24 hours apart (Day-1 and Day-2). At the end of Day-1, an eccentric exercise is performed in order to to induce delayed onset muscle soreness on the external rotators of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and free from any pain specific to the upper limbs and/or in general.

Exclusion Criteria:

* Previous history of chronic pain.
* Any systemic diseases or regional pathology which can interfere with the outcome measures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with no acute pain, chronic pain or other medical disorders relevant to this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in temperature of pixels on the upper extremity: infrared thermography | Day-1 (baseline assessment, pre exercise before painful stimulus), Day-1 (baseline assessment, pre exercise after painful stimulus), Day-2 (24 hours post-exercise before painful stimulus), Day-2 (24 hours post-exercise after painful stimulus)
  A thermography image of the upper extremity of the body will be taken on both days of assessment before and after applying a painful stimulus. Changes in colour pixels will be analysed to determine temperature changes.

SECONDARY OUTCOMES:
Changes in Pressure Pain Thresholds: pressure algometry | Day-1 (baseline assessment, pre exercise before painful stimulus), Day-2 (24 hours post-exercise before painful stimulus)
  Changes in pressure pain thresholds will be determined with pressure algometry over the infraspinatus muscle. Pressure Pain Threshold is defined as the exact time point where the pressure is first being perceived as painful.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, PhD, Study Director — Universidad San Jorge

IPD SHARING:
Plan to Share IPD: No
There are currently no plan on sharing data from this study with other researchers.